CLINICAL TRIAL: NCT04982848
Title: A Prospective, Single-arm, Open-label, Non-interventional, Multi-centre, Post Marketing Surveillance (PMS) Study of Talzenna(Registered)
Brief Title: Korea Post Marketing Surveillance (PMS) Study of Talzenna®
Status: Not yet recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3441038; Talzenna PMS (Other: Alias Study Number)
Record Dates: First submitted 2021-07-14; First posted 2021-07-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Neoplasms
Keywords: gBRCA
MeSH Terms: conditions — Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Talzenna treated group: Talzenna treated gBRCA Breast cancer patients in the real world setting in Korea
  Interventions: Drug: Talzenna

INTERVENTIONS:
Drug: Talzenna — Talzenna treatment under Korea regulatory approval indication/dosage

SUMMARY:
Talzenna will be approved for the treatment of gBRCA advanced breast cancer in Korea. In accordance with the Standards for Re-examination of New Drug, it is required to conduct a PMS. Post marketing surveillance is required to determine any problems or questions associated with Talzenna after marketing in Korea, with regard to the following clauses under conditions of general clinical practice. Therefore, through this study, effectiveness and safety of Talzenna will be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled to start treatment with Talzenna® based on the clinical judgment of their treating physician as specified in the Korean-Prescribing information (local label)
2. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. Patients with known hypersensitivity to Talzenna®, or to any of the excipients.
2. Breastfeeding
3. Any patients (or a legally acceptable representative) who does not agree that Pfizer and companies working with Pfizer use his/her information.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Talzenna® is indicated as monotherapy for the treatment of adult patients with breast cancer susceptibility gene (BRCA) mutated human epidermal growth factor receptor 2 (HER2)-negative locally advanced or metastatic breast cancer who have been treated with chemotherapy in the neoadjuvant, adjuvant, or advanced setting.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2027-06-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events categorized according to physical organ and disease/symptom | From date of randomization until the 28 calendar days following the last administration of a drug under study
  It is non-interventional, observational study in the real world setting. Adverse events will be captured in the real world clinical practice.

SECONDARY OUTCOMES:
Overal response (Effectiveness outcome) by Response Evaluation Criteria In Solid Tumors (RECIST) critera | through study completion, an expected average of 8 months
  It is non-interventional, observational study in the real world setting. Response evaluation will be assessed based on the real world clinical practice

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.